CLINICAL TRIAL: NCT05628753
Title: Lung Ultrasound as a Predictor for Successful Extubation in Preterm Infants
Acronym: LUSE
Status: Completed | Type: Observational
Sponsor: Royal University Hospital, Saskatoon (Other)
Responsible Party: Sponsor
Other Study IDs: Bio ID 1451
Record Dates: First submitted 2022-11-16; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: no Conditions
Keywords: Lung ultrasound; Prematurity; RDS; Mechanical ventilation; Extubation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound (LUS) — LUS performed 30 mins prior to and 120 minutes after planned extubation with a linear high frequency probe longitudinal approach was used in all three zones Repeated third scan will be done prior to re-intubation (if required) The ultrasound total execution cut-off time expected to be less than 5 minutes

SUMMARY:
unit (NICU); however prolonged MV is known to be associated with serious complications including ventilator associated pneumonia, blood stream infections, bronchopulmonary dysplasia (BPD) and periventricular leukomalacia. At the same time, extubation failure increases morbidities and mortality. Hatch et al (2016) in their prospective study on 162 infants described adverse events in 40% of intubations and severe complications including need for CPR in 9%. Reintubations are frequently associated with hypoxemia, bradycardia, fluctuations in blood pressures and cerebral perfusion. Each intubation attempt increases the risk of traumatic injury to the upper airway, lung atelectasis and infections. Thus, there is a clear need to establish objective criteria that would help avoid extubation failure and the need for reintubation.

In recent years, a new imaging application has been introduced in neonatal practice-lung ultrasound (LUS), an accurate and reliable technique for the lung evaluation. LUS is safe, non-ionizing, easy to operate, and low-cost tool. The evaluation of lungs is performed in real-time, on the bedside and without anesthetic drugs. Lung aeration could be assessed in dynamics without extra radiation to the infant. Ultrasound findings combined with clinical information could be used for the prognosis of successful extubation in premature infants.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is a widely used therapeutic resource in neonatal intensive care unit (NICU); however prolonged MV is known to be associated with serious complications including ventilator associated pneumonia, blood stream infections, bronchopulmonary dysplasia (BPD) and periventricular leukomalacia. At the same time, extubation failure increases morbidities and mortality. Hatch et al (2016) in their prospective study on 162 infants described adverse events in 40% of intubations and severe complications including need for CPR in 9%. Reintubations are frequently associated with hypoxemia, bradycardia, fluctuations in blood pressures and cerebral perfusion. Each intubation attempt increases the risk of traumatic injury to the upper airway, lung atelectasis and infections. Thus, there is a clear need to establish objective criteria that would help avoid extubation failure and the need for reintubation.

Currently used criteria for extubation are subjective and based on clinical evaluation, chest radiograph findings, amount of ventilatory support and arterial blood gas (ABG) parameters. An accurate bedside test for extubation readiness in preterm infants born is even more important as this population is more susceptible to the complications of re-intubation. There are several studies that showed that reintubation after elective extubation is independently associated with increased likelihood of death and BPD in extremely preterm infants. The greatest risks are attributable to reintubation within the first 48 hours post-extubation.

Several studies have shown that a low lung volume and small chest radiograph lung area after extubation could predict extubation failure. Infants who have a low lung volume after extubation may have an unfavourable balance between respiratory muscle strength and respiratory load. Ideally, these infants should be identified before removal of the endotracheal tube.

In recent years, a new imaging application has been introduced in neonatal practice-lung ultrasound (LUS), an accurate and reliable technique for the lung evaluation. LUS is safe, non-ionizing, easy to operate, and low-cost tool. The evaluation of lungs is performed in real-time, on the bedside and without anesthetic drugs. Lung aeration could be assessed in dynamics without extra radiation to the infant. Ultrasound findings combined with clinical information could be used for the prognosis of successful extubation in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Invasively ventilated infants born at less than 32 weeks of gestational age were included at the time of their first extubation

Exclusion Criteria:

* infants born after 32 weeks of gestational age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Invasively ventilated infants born before 32 weeks of gestational age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
lung aeration before and after extubation by comparing LUS indexes | 30 minutes
re-intubation within 12, 36 or 72 hours | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided